CLINICAL TRIAL: NCT00002202
Title: A Phase III Trial to Compare the Safety and Antiviral Efficacy of 141W94 With Indinavir in Combination With Nucleoside Reverse Transcriptase Inhibitor (NRTI) Therapy, in NRTI-Experienced, Protease Inhibitor (PI)-Naive, HIV-1-Infected Patients.
Brief Title: A Comparison of 141W94 and Indinavir in HIV-Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 264E; PROA/B3006
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-11

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; HIV Protease Inhibitors; Indinavir; RNA, Viral; VX 478; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; amprenavir

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Amprenavir

SUMMARY:
The purpose of this study is to see if 141W94 is as safe and effective as indinavir when used with nucleoside reverse transcriptase inhibitors (NRTIs) for 48 weeks. This study also examines what effect other drugs have on how the body handles 141W94.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented HIV infection.
* HIV RNA >= 400 copies/ml within 14 days prior to randomized study drug administration.
* No active AIDS-defining opportunistic infection or disease.
* Signed, informed consent from parent or legal guardian of patients less than 18 years of age.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Unlikely to complete the randomized dosing period.
* Malabsorption syndrome or other gastrointestinal dysfunction that might interfere with drug absorption or ability to take oral medications.
* Serious medical conditions (e.g., diabetes, cardiac dysfunction, hepatitis) that would compromise patient safety.

Concurrent Medication:

Excluded:

* Cytotoxic chemotherapeutic agents (except local treatment for Kaposi's sarcoma).
* Investigational treatments (treatment through Treatment IND or expanded-access programs are evaluated individually).
* Immunomodulating agents such as systemic, high-dose corticosteroids, interleukins, or interferons.
* Terfenadine, astemizole, cisapride, triazolam, midazolam, and ergotamine/dihydroergotamine-containing regimens.

Concurrent Treatment:

Excluded:

Radiation therapy (except local treatment for Kaposi's sarcoma).

Patients with the following prior conditions are excluded:

Clinically relevant pancreatitis or hepatitis within the last 6 months.

Prior Medication:

Excluded:

* Cytotoxic chemotherapeutic agents within 30 days of study drug administration (except local treatment for Kaposi's sarcoma).
* Protease inhibitor therapy.
* Dose of vaccine through an investigational HIV vaccine trial within the 3 months prior to study drug administration.
* Immunomodulating agents such as systemic, high-dose corticosteroids, interleukins, or interferons within 30 days of study drug administration.

Prior Treatment:

Excluded:

Radiation therapy within 30 days prior to study drug administration (except local treatment for Kaposi's sarcoma).

Risk Behavior:

Excluded:

Current alcohol or illicit drug use that may interfere with drug absorption or ability to take oral medication.

Required:

NRTI therapy at day of entry and up to screening.

Required:

>= 12 weeks of NRTI therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - East Bay AIDS Ctr, Berkeley, California
  - AIDS Healthcare Foundation, Los Angeles, California
  - Saint Francis Mem Hosp, San Francisco, California
  - ViRx Inc, San Francisco, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Whitman Walker Clinic Inc, Washington D.C., District of Columbia
  - CRI of South Florida, Coral Gables, Florida
  - Community Research Initiative of Central Florida, Maitland, Florida
  - Univ of Miami Dept of Medicine, Miami, Florida
  - Northwestern Univ Med School, Chicago, Illinois
  - Tulane Univ Med School, New Orleans, Louisiana
  - Boston Med Ctr / Evans - 556, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - Community Research Initiative on AIDS, New York, New York
  - Harlem Hosp, New York, New York
  - The Nalle Clinic / Clinical Research Dept, Charlotte, North Carolina
  - Med College of Ohio / Division of Infectious Diseases, Toledo, Ohio
  - The Research and Education Group, Portland, Oregon
  - Methodist Hosp, Memphis, Tennessee
  - Community Oriented Primary Care, Dallas, Texas
  - Univ of Texas Med Branch, Galveston, Texas
  - Baylor College of Medicine / Dept of Medicine, Houston, Texas
  - Hampton Roads Med Specialists, Hampton, Virginia